CLINICAL TRIAL: NCT07031609
Title: Spastik Hemiparetik Serebral Palsili Bireylerde Robotik Destekli Yürüyüş Eğitimi, Hidroterapi ve Konvansiyoel Fizyoterapi Yöntemlerinin Kas Kuvveti, Denge, Fonksiyonel Mobilite ve Ruhsal Uyum Üzerindeki Etkileri
Brief Title: Effects of Robotic Gait, Hydrotherapy, and Conventional Physiotherapy in Spastic Hemiparetic CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Collaborators: Kayseri University (Other)
Responsible Party: Principal Investigator, Ozge Baykan Copuroglu, Asst. Prof., Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KayseriUniversity
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy
Keywords: Spastic Hemiparetic Cerebral Palsy; Robot-Assisted Gait Training; Hydrotherapy; Conventional Physiotherapy; Pediatric Rehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with a parallel assignment model. Participants will be randomly allocated into three parallel intervention groups: (1) robot-assisted gait training, (2) hydrotherapy, and (3) conventional physiotherapy. Each group will receive two sessions per week for six weeks. The interventions will be administered independently, with no crossover between groups. Outcome measures will be assessed at baseline and after the six-week intervention period.
Masking Description: No masking will be implemented in this study. All participants, care providers, investigators, and outcome assessors will be aware of the assigned interventions due to the nature of the treatment protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot-Assisted Gait Training Group (Experimental): Participants in this arm will receive robot-assisted gait training using the Lokomat device for 40 minutes, twice a week, over a 6-week period. The intervention aims to improve lower limb muscle strength, balance, and mobility.
  Interventions: Behavioral: Robot-assisted gait training using Lokomat
- Hydrotherapy Group (Experimental): Participants will undergo supervised aquatic exercises in a therapeutic pool for 40 minutes, twice a week, for 6 weeks. The exercises are designed to enhance strength, coordination, and balance in children with spastic hemiparetic cerebral palsy.
  Interventions: Behavioral: Hydrotherapy
- Conventional Physiotherapy Group (Experimental): This group will receive conventional physiotherapy consisting of electrotherapy (faradic stimulation), passive and active range of motion exercises, gait training, and positioning techniques. Sessions last 40 minutes, twice a week, for 6 weeks.
  Interventions: Behavioral: Conventional Physiotherapy

INTERVENTIONS:
Behavioral: Robot-assisted gait training using Lokomat — This intervention involves robotic-assisted gait training with the Lokomat device. Sessions will last 40 minutes, twice a week for 6 weeks. The intervention targets lower extremity motor function in children with spastic hemiparetic cerebral palsy. The robotic system provides adjustable support and real-time feedback to improve gait patterns and mobility.
  Other Names: Lokomat-based gait rehabilitation
  Arms: Robot-Assisted Gait Training Group
Behavioral: Hydrotherapy — Participants will engage in supervised aquatic therapy including structured exercises in a therapeutic pool. Each session lasts 40 minutes, twice a week, for 6 weeks. Exercises include water walking, floating resistance training, jumping, and balance activities designed for children with spastic hemiparetic cerebral palsy to improve strength, coordination, and functional mobility.
  Other Names: Aquatic exercise program; Water-based physiotherapy
  Arms: Hydrotherapy Group
Behavioral: Conventional Physiotherapy — This intervention includes 20 minutes of faradic electrical stimulation and 20 minutes of therapeutic exercises such as stretching, positioning, range of motion, and gait training. Administered twice a week for 6 weeks. The protocol aims to support neuromuscular activation and improve gait and mobility in children with spastic hemiparetic cerebral palsy.
  Other Names: Standard conventional physiotherapy; Traditional physiotherapy
  Arms: Conventional Physiotherapy Group

SUMMARY:
This study aims to evaluate the effects of three different physiotherapy approaches-robot-assisted gait training, hydrotherapy, and conventional physiotherapy-on muscle strength, balance, functional mobility, and psychological adjustment in children diagnosed with spastic hemiparetic cerebral palsy. A total of 45 ambulatory children aged 5 to 15 years will be randomly assigned to one of the three intervention groups. All participants will receive therapy twice a week for six weeks.

Muscle strength will be assessed using a handheld dynamometer, balance with the Pediatric Balance Scale, mobility with the Timed Up and Go test, and psychological adjustment with a standardized behavioral checklist. The study will help determine which therapeutic approach provides the most benefit in improving physical function and emotional well-being. Results may guide healthcare providers and families in selecting the most effective rehabilitation method for children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 5 and 15 years
* Diagnosed with spastic hemiparetic cerebral palsy
* Classified as Level I or II on the Gross Motor Function Classification System (GMFCS)
* Able to follow simple instructions and participate in therapy sessions
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Severe cognitive or mental impairment that interferes with communication
* Lower extremity joint contractures preventing use of robotic gait device
* Uncontrolled cardiac disease
* Active infection at the time of intervention
* Open skin lesions on the legs or trunk
* Inability to properly fit orthoses required for therapy
* Withdrawal of consent by the child or parent/guardian
* Failure to complete the assessment tests
* New illness or surgical intervention during the study period

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | Baseline and Week 6
  Change in lower extremity muscle strength measured by hand-held dynamometer (MicroFET® 2) at baseline and after 6 weeks of intervention.
Balance | Baseline and Week 6
  Change in balance performance assessed by Pediatric Balance Scale (PBS).
Functional Mobility | Baseline and Week 6
  Change in mobility measured using the Timed Up and Go (TUG) test.

SECONDARY OUTCOMES:
Psychological Adjustment | Baseline and Week 6
  Change in psychosocial adjustment scores based on the Hacettepe Psychological Adjustment Scale for Children (parent-rated).
Treatment Tolerance and Adherence | Ongoing through 6 weeks
  Number of completed sessions out of 12 scheduled sessions during the 6-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686